CLINICAL TRIAL: NCT04355468
Title: Opioid-free Anaesthesia Effectiveness in Thoracic Surgery - Objective Measurement With a Skin Conductance Algesimeter: a Randomized Controlled Trial
Brief Title: Opioid Free Anesthesia in Thoracic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Silesia (Other)
Responsible Party: Principal Investigator, Piotr Palaczyński, Principal Investigator, Medical University of Silesia
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: OPA-1
Record Dates: First submitted 2020-04-18; First posted 2020-04-21 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-10

CONDITIONS: Thoracic Surgery; Analgesics, Opioid; Anesthesia, Conduction

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): General anesthesia was induced with midazolam 0.1 mg∙kg-1, propofol 2 mg∙kg-1, and cisatracurium 0.15 mg∙kg-1. The patients were intubated with a left-sided double-lumen tube in adequate size and positioned laterally. Anesthesia was maintained with 1 minimum alveolar concentration (MAC) sevoflurane. The patients awoke from anesthesia in a post-anesthesia care unit, and were extubated after the administration of adequate doses of atropine and neostigmine as required. After surgery, if a patient complained of pain then she/he was given i.v. oxycodone by an anesthetist before commencing the patient controlled analgesia (PCA). This dose was titrated to achieve adequate analgesia. Each patient then commenced PCA. The PCA solution was oxycodone (1mgml-1) and the PCA was programmed to allow a self-administered bolus dose of 1mg oxycodone with a lockout time of 5 min. Additionally, patients were given 1 g intravenous paracetamol every 6 h and 100mg of intravenous ketoprofen every 12 h.
  Interventions: Drug: Opioid Anesthesia
- Opioid Free Aneasthesia group (Experimental): General anesthesia was induced with midazolam 0.1 mg∙kg-1, propofol 2 mg∙kg-1, and cisatracurium 0.15 mg∙kg-1. The patients were intubated with a left-sided double-lumen tube in adequate size and positioned laterally. Anesthesia was maintained with 1 minimum alveolar concentration (MAC) sevoflurane. The patients awoke from anesthesia in a post-anesthesia care unit, and were extubated after the administration of adequate doses of atropine and neostigmine as required. After surgery, if a patient complained of pain then she/he was given i.v. oxycodone by an anesthetist before commencing the patient controlled analgesia (PCA). This dose was titrated to achieve adequate analgesia. Each patient then commenced PCA. The PCA solution was oxycodone (1mgml-1) and the PCA was programmed to allow a self-administered bolus dose of 1mg oxycodone with a lockout time of 5 min. Additionally, patients were given 1 g intravenous paracetamol every 6 h and 100mg of intravenous ketoprofen every 12 h.
  Interventions: Drug: Opioid Free Anaesthesia

INTERVENTIONS:
Drug: Opioid Anesthesia — Intraoperatively, fentanyl in fractional doses of 1-3 µg∙kg-1 were applied if the heart rate (HR; Heart Rate) or mean blood pressure (MBP; Mean Blood Pressure) increased by more than 20% above the baseline value obtained just before surgery commencement.
  Arms: Control group
Drug: Opioid Free Anaesthesia — Before the induction of general anesthesia, a single-shot thoracic paravertebral block (ThPVB) was performed at the Th3-Th4 level. An insulated needle was used, connected to a peripheral nerve stimulator. 0.5% bupivacaine (0.3 ml∙kg-1) was then injected after a negative aspiration test. The efficacy of the blockade was checked after 20 min on both sides of the thorax with a plastic ampoule of saline. A difference in the sensation of cold between the sides of the thorax was assumed to indicate an effective block. Afterwards a continuous intravenous infusion of lidocaine and ketamine was started:
  1. immediately after anesthesia induction, lidocaine was administered as an i.v. bolus at a dose of 1.5 mg∙kg-1 and ketamine in an i.v. bolus of 0.35 mg∙kg-1;
  2. followed by an infusion of lidocaine 2.0 mg∙kg-1∙h-1 for 2 hours, continued at a dose of 1.2 mg∙kg-1∙h-1, and ketamine infusion 0.2 mg∙kg-1∙h-1 for 2 hours, continued at a dose of 0.12 mg∙kg-1∙h-1.
  Arms: Opioid Free Aneasthesia group

SUMMARY:
Proper assessment of pain and adequate analgesia in thoracic surgery is a challenging issue for medical practitioners. Basic aspects of thoracic anaesthesia are general anesthesia, intubation with double lumen tube and separation of lung ventilation, however proper analgesia needs to be standardized. Role of opioids in this clinical setting is reduced due to high risk of respiratory system complications. Instead, use of opioid free anaesthesia and regional anaesthesia is proposed. The aim of this study is to compare the use of opioid anaesthesia with opioid free anaesthesia and paravertebral block.

ELIGIBILITY:
Inclusion Criteria:

* body mass index between 19-30 kg/m2,
* American Society of Anesthesiology (ASA) physical status between 1 and 3

Exclusion Criteria:

* lack of consent
* significant coagulopathy,
* contraindication to drugs used in protocol
* history of chronic pain,
* chest wall neoplastic invasion,
* previous thoracic spine surgery,
* mental state preventing from effective use of PCA device,
* renal failure (GFR <60 ml/min/1,73 m2)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Intraoperative pain related stress [oscillations per second] | Period before induction of anaesthesia to termination of anaesthesia
  During general anesthesia the pain-related stress was assessed using a method of skin conductance fluctuations. The measurement was based on changes in skin conductance that arise under the influence of a pain stimulus.
Intraoperative opioid usage [mg] | Intraoperative period
  Intraoperative usage of opioids was noted.
Intraoperative arterial blood pressure [mmHg] | Intraoperative period
  Non-invasive arterial blood pressure was recorded every 5 minutes during operation.
Intraoperative heart rate [bpm] | Intraoperative period
  Heart rate was recorded every 5 minutes during operation.

SECONDARY OUTCOMES:
Overall postoperative analgesia satisfaction | 48 hours
  Overall analgesia satisfaction was recorded at 24 and 48 postoperative hours with Likert scale. The points in Likert scale were assigned as below:
  1. Very satisfied.
  2. Satisfied.
  3. Neither satisfied nor dissatisfied.
  4. Dissatisfied.
  5. Very dissatisfied.
Postoperative pain intensity (VAS) | 48 hours
  Pain intensity at rest was recorded with Visual Analogue Scale (VAS) at 0, 1, 2, 4, 8, 12, 18, 24, 30, 36, 42, 48 postoperative hours. Patient pointed intensity of symptoms on a 10cm ruler, where 0cm corresponded to no pain and 10cm corresponded to the strongest possible pain.
Postoperative pain intensity (PHHPS) | 48 hours
  Pain intensity at rest was recorded with Prince Henry Hospital Pain Score (PHHPS) at 0, 1, 2, 4, 8, 12, 18, 24, 30, 36, 42, 48 postoperative hours. The points in PHHPS score were assigned as below:
  0. No pain during coughing.
  1. Pain during coughing.
  2. Pain during breathing.
  3. Constant light pain.
  4. Constant strong pain.
Postoperative arterial blood pressure [mmHg] | 48 hours
  Non-invasive arterial blood pressure was recorded at 0, 1, 2, 4, 8, 12, 18, 24, 30, 36, 42, 48 postoperative hours.
Postoperative heart rate [bmp] | 48 hours
  Heart rate was recorded at 0, 1, 2, 4, 8, 12, 18, 24, 30, 36, 42, 48 postoperative hours.
Postoperative sedation level | 48 hours
  Sedation level was was recorded at 0, 1, 2, 4, 8, 12, 18, 24, 30, 36, 42, 48 postoperative hours with Ramsay scale. The points in Ramsay scale were assigned as below:
  1. Patient is anxious and agitated or restless, or both.
  2. Patient is co-operative, oriented, and tranquil.
  3. Patient responds to commands only.
  4. Patient exhibits brisk response to light glabellar tap or loud auditory stimulus.
  5. Patient exhibits a sluggish response to light glabellar tap or loud auditory stimulus.
  6. Patient exhibits no response.
Postoperative analgesic requirement [mg] | 48 hours
  Analgesic requirement was recorded at 0, 1, 2, 4, 8, 12, 18, 24, 30, 36, 42, 48 postoperative hours.

CONTACTS AND LOCATIONS:
Locations (1):
- Samodzielny Publiczny Szpital Kliniczny nr 1, Zabrze, Silesian Voivodeship, Poland